CLINICAL TRIAL: NCT05541471
Title: A Phase 1, Open-label Study to Evaluate Pharmacokinetic Drug-drug Interactions Between VX-548 and Midazolam and Digoxin in Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetic Drug-drug Interactions Between VX-548, Midazolam, and Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: VX21-548-010
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Midazolam; Digoxin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Participants will receive a single dose of midazolam and digoxin on Day 1 in dosing period 1 followed by VX-548 every 12 hours (q12h) on Days 6 through 23 in dosing period 2. On Day 19, single doses of midazolam and digoxin will be administered with the morning dose of VX-548.
  Interventions: Drug: VX-548; Drug: Midazolam; Drug: Digoxin

INTERVENTIONS:
Drug: VX-548 — Tablets for oral administration.
  Other Names: Suzetrigine
Drug: Midazolam — Syrup for oral administration.
Drug: Digoxin — Tablets for oral administration.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of midazolam and digoxin in the absence and presence of VX-548.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (Kg/m^2)
* A total body weight greater than (>) 50 kilogram (kg)
* Females of non-childbearing potential

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 5 days before the first dose of study drug
* Any condition possibly affecting drug absorption
* History of cardiovascular disease, cardiac dysrhythmias or central nervous system disease
* Hypersensitivity to midazolam, other benzodiazepines, or digoxin

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Midazolam in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 24 hours post midazolam dose
Maximum Observed Plasma Concentration (Cmax) of Digoxin in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 120 hours post digoxin dose
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of Midazolam in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 24 hours post midazolam dose
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of Digoxin in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 120 hours post digoxin dose
Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of Midazolam in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 24 hours post midazolam dose
Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of Digoxin in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 120 hours post digoxin dose

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of 1-hydroxy-Midazolam in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 24 hours post midazolam dose
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of 1-hydroxy-Midazolam in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 24 hours post midazolam dose
Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of 1-hydroxy-Midazolam in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 24 hours post midazolam dose
Renal Clearance (CLr) of Digoxin as Determined by Urine Analysis in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 120 hours post digoxin dose
Fraction of Systematically Available Digoxin Dose Excreted Unchanged (fe) in Urine in the Absence and Presence of VX-548 | Days 1 and 19: Pre-dose up to 120 hours post digoxin dose
Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 39
Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Pre-dose up to Day 39

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore - Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing